CLINICAL TRIAL: NCT03186989
Title: A Randomized, Double-Blind, Placebo-Controlled Study, Followed by an Open-Label Extension, to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Doses of Intrathecally Administered ISIS 814907 in Patients With Mild Alzheimer's Disease
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IONIS-MAPTRx in Patients With Mild Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ISIS 814907-CS1; NL60032.000.16 (Other: CCMO); 2016-002713-22 (EudraCT Number)
Record Dates: First submitted 2017-06-06; First posted 2017-06-14 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Mild Alzheimer's Disease
Keywords: Mild Alzheimer's Disease; ISIS 814907; Memory Loss; Alzheimers; MAPT; Tau
MeSH Terms: conditions — Memory Disorders; Pick Disease of the Brain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (11):
- Part 1: Cohort A: ISIS 814907 10 mg (Experimental): Participants received 10 milligrams (mg) ISIS 814907 diluted in 20 milliliters (mL) artificial cerebrospinal fluid (CSF), intrathecally, every four weeks (Q4W) on Days 1, 29, 57, and 85 in Part 1 of the study.
  Interventions: Drug: IONIS MAPTRx
- Part 1: Cohort B: ISIS 814907 30 mg (Experimental): Participants received 30 mg ISIS 814907 diluted in 20 mL in artificial CSF, intrathecally, Q4W on Days 1, 29, 57, and 85 in Part 1 of the study.
  Interventions: Drug: IONIS MAPTRx
- Part 1: Cohort C: ISIS 814907 60 mg (Experimental): Participants received 60 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, Q4W on Days 1, 29, 57, and 85 in Part 1 of the study.
  Interventions: Drug: IONIS MAPTRx
- Part 1: Cohort D: ISIS 814907 115 mg (Experimental): Participants received 115 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, every 12 weeks (Q12W) on Days 1 and 85 in Part 1 of the study.
  Interventions: Drug: IONIS MAPTRx
- Part 1: Pooled Placebo (Placebo Comparator): Participants received 20 mL artificial CSF, intrathecally, as placebo on Days 1, 29, 57, and 85 for the 4-dose regimens, or on Days 1 and 85 for the 2-dose regimens in Part 1 of the study.
  Interventions: Other: Placebo
- Part 2: Late Start Cohort A + Cohort B + Cohort C + ISIS 814907 60 mg (Experimental): Participants from MAD Cohorts A, B, C that were placebo-treated, received 60 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, Q12W on Days 1, 85, 169, 253, and 337 in Part 2 of the study.
  Interventions: Drug: IONIS MAPTRx
- Part 2: Late Start Cohort D + ISIS 814907 115 mg (Experimental): Participants from MAD Cohort D that were placebo-treated, received 115 mg ISIS 814907 diluted up in 20 mL artificial CSF, intrathecally, Q12W on Days 1, 85, 169, 253, and 337 in Part 2 of the study.
  Interventions: Drug: IONIS MAPTRx
- Part 2: Early Start Cohort A + ISIS 814907 60 mg (Experimental): Participants from MAD Cohort A that were ISIS 814907 10 mg -treated, received 60 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, Q12W on Days 1, 85, 169, 253, and 337 in Part 2 of the study.
  Interventions: Drug: IONIS MAPTRx
- Part 2: Early Start Cohort B + ISIS 814907 60 mg (Experimental): Participants from MAD Cohort B that were ISIS 814907 30 mg-treated, received 60 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, Q12W on Days 1, 85, 169, 253, and 337 in Part 2 of the study.
  Interventions: Drug: IONIS MAPTRx
- Part 2: Early Start Cohort C + ISIS 814907 60 mg (Experimental): Participants from MAD Cohort C that were ISIS 814907 60 mg-treated, received 60 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, Q12W on Days 1, 85, 169, 253, and 337 in Part 2 of the study.
  Interventions: Drug: IONIS MAPTRx
- Part 2: Early Start Cohort D + ISIS 814907 115 mg (Experimental): Participants from MAD Cohort D that were ISIS 814907 115 mg-treated, received 115 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, Q12W on Days 1, 85, 169, 253, and 337 in Part 2 of the study.
  Interventions: Drug: IONIS MAPTRx

INTERVENTIONS:
Drug: IONIS MAPTRx — IONIS MAPTRx injections.
  Other Names: ISIS 814907
  Arms: Part 1: Cohort A: ISIS 814907 10 mg; Part 1: Cohort B: ISIS 814907 30 mg; Part 1: Cohort C: ISIS 814907 60 mg; Part 1: Cohort D: ISIS 814907 115 mg; Part 2: Early Start Cohort A + ISIS 814907 60 mg; Part 2: Early Start Cohort B + ISIS 814907 60 mg; Part 2: Early Start Cohort C + ISIS 814907 60 mg; Part 2: Early Start Cohort D + ISIS 814907 115 mg; Part 2: Late Start Cohort A + Cohort B + Cohort C + ISIS 814907 60 mg; Part 2: Late Start Cohort D + ISIS 814907 115 mg
Other: Placebo — Artificial CSF injections.
  Arms: Part 1: Pooled Placebo

SUMMARY:
The purpose of this study was to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of IONIS-MAPTRx in patients with Mild Alzheimer's Disease.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled study in 46 participants, followed by an Open-Label Extension. This study consisted of two parts:

Part 1: a randomized, double-blind, placebo-controlled multiple ascending dose period in participants with Mild Alzheimer's Disease, followed by Part 2: the open-label, long-term extension period.

ELIGIBILITY:
Inclusion Criteria for Part 1:

* Males or females aged 50-74 years, inclusive, at the time of informed consent
* Diagnosed with mild Alzheimers disease, including CSF biomarkers consistent with this diagnosis
* Body Mass Index BMI ≥ 18 and ≤ 35 kg/m2 and total body weight > 50 kg (110 lbs)
* Able and willing to meet all study requirements, including toleration for MRI scans, blood draws and lumbar punctures, travel to Study Center and participation in all procedures and measurements at study visits
* Have a trial partner who is reliable, competent and at least 18 years of age, is willing to accompany the patient to select trial visits and to be available to the Study Center by phone if needed
* Reside within 4 hours travel of the Study Center

Exclusion Criteria for Part 1:

* Treatment with another Study Drug, biological agent, or device within one-month of Screening or 5 half-lives of investigational agent, whichever is longer
* Clinically significant medical condition which would make the patient unsuitable for inclusion or could interfere with the patient participating in or completing the study
* Use of a disallowed CNS-active or antipsychotic medication within 4 weeks prior to Screening punctures

Inclusion Criteria for Part 2:

* Must have completed the Treatment Evaluation and Post-Treatment Periods in Part 1

Exclusion Criteria for Part 2 (only applicable to participants in Cohorts A and B, as participants from Cohorts C and D will seamlessly transition to Part 2):

* Treatment with another Study Drug, biological agent, or device within one-month of Screening or 5 half-lives of investigational agent, whichever is longer
* Clinically significant medical condition which would make the patient unsuitable for inclusion or could interfere with the patient participating in or completing the study
* Use of a disallowed CNS-active or antipsychotic medication within 4 weeks prior to Screening punctures

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Montreal Neurological Hospital, Montreal, Canada
- Clinical Research Services Turku CRST, Turku, Finland
- Germany (4):
  - St Josef Hospital, Bochum
  - Deutsches Zentrum für Neurodegenerative Erkrankungen (DZNE), Bonn
  - MVZ Mittweida Gbr, Mittweida
  - Universittsklinikum Ulm, Ulm
- Netherlands (2):
  - VU University Medical Center, Amsterdam
  - QPS Netherlands BV, Groningen
- Sweden (2):
  - Minnesmottagningen, Mölndal
  - Karolinska University Hospital Huddinge, Stockholm
- United Kingdom (3):
  - Royal Liverpool University Hospital, Liverpool
  - University College London Hospitals NHS Foundation Trust, London
  - Sheffield Institute for Translational Neuroscience (SITraN), Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lane RM, Darreh-Shori T, Junge C, Li D, Yang Q, Edwards AL, Graham DL, Moore K, Mummery CJ. Onset of Alzheimer disease in apolipoprotein varepsilon4 carriers is earlier in butyrylcholinesterase K variant carriers. BMC Neurol. 2024 Apr 9;24(1):116. doi: 10.1186/s12883-024-03611-5. PMID 38594621
- [Derived] Edwards AL, Collins JA, Junge C, Kordasiewicz H, Mignon L, Wu S, Li Y, Lin L, DuBois J, Hutchison RM, Ziogas N, Shulman M, Martarello L, Graham D, Lane R, Budd Haeberlein S, Beaver J. Exploratory Tau Biomarker Results From a Multiple Ascending-Dose Study of BIIB080 in Alzheimer Disease: A Randomized Clinical Trial. JAMA Neurol. 2023 Dec 1;80(12):1344-1352. doi: 10.1001/jamaneurol.2023.3861. PMID 37902726
- [Derived] Mummery CJ, Borjesson-Hanson A, Blackburn DJ, Vijverberg EGB, De Deyn PP, Ducharme S, Jonsson M, Schneider A, Rinne JO, Ludolph AC, Bodenschatz R, Kordasiewicz H, Swayze EE, Fitzsimmons B, Mignon L, Moore KM, Yun C, Baumann T, Li D, Norris DA, Crean R, Graham DL, Huang E, Ratti E, Bennett CF, Junge C, Lane RM. Tau-targeting antisense oligonucleotide MAPTRx in mild Alzheimer's disease: a phase 1b, randomized, placebo-controlled trial. Nat Med. 2023 Jun;29(6):1437-1447. doi: 10.1038/s41591-023-02326-3. Epub 2023 Apr 24. PMID 37095250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 investigative sites in the Germany, United Kingdom, the Netherlands, Sweden, Canada, and Finland from 23 August 2017 to 12 May 2022.
Pre-assignment Details: A total of 102 participants were screened and 46 participants with mild Alzheimer's disease were enrolled and randomized to receive ISIS 814907 or placebo in Part 1 (multiple ascending dose [MAD]). This study consists of two parts i.e., Part 1: MAD and Part 2: long-term extension (LTE). Out of 46 participants enrolled in Part 1, 33 participants who met the pre-specified eligibility criteria transitioned into Part 2.
Groups:
- Part 1: Cohort A: ISIS 814907 10 mg: Participants received 10 milligrams (mg) ISIS 814907 diluted in 20 millilitres (mL) artificial cerebrospinal fluid (CSF), intrathecally, every four weeks (Q4W) on Days 1, 29, 57, and 85 in Part 1 of the study.
Period: Part 1: MAD (Day 1 up to Week 36)
Arm/Group | Part 1: Cohort A: ISIS 814907 10 mg | Part 1: Cohort B: ISIS 814907 30 mg | Part 1: Cohort C: ISIS 814907 60 mg | Part 1: Cohort D: ISIS 814907 115 mg | Part 1: Pooled Placebo | Part 2: Late Start Cohort A + Cohort B + Cohort C + ISIS 814907 60 mg | Part 2: Late Start Cohort D + ISIS 814907 115 mg | Part 2: Early Start Cohort A + ISIS 814907 60 mg | Part 2: Early Start Cohort B + ISIS 814907 60 mg | Part 2: Early Start Cohort C + ISIS 814907 60 mg | Part 2: Early Start Cohort D + ISIS 814907 115 mg
Started | 6 | 6 | 9 | 13 | 12 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 6 | 8 | 12 | 11 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Voluntary Withdrawal | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: LTE (Week 37 to Week 101)
Arm/Group | Part 1: Cohort A: ISIS 814907 10 mg | Part 1: Cohort B: ISIS 814907 30 mg | Part 1: Cohort C: ISIS 814907 60 mg | Part 1: Cohort D: ISIS 814907 115 mg | Part 1: Pooled Placebo | Part 2: Late Start Cohort A + Cohort B + Cohort C + ISIS 814907 60 mg | Part 2: Late Start Cohort D + ISIS 814907 115 mg | Part 2: Early Start Cohort A + ISIS 814907 60 mg | Part 2: Early Start Cohort B + ISIS 814907 60 mg | Part 2: Early Start Cohort C + ISIS 814907 60 mg | Part 2: Early Start Cohort D + ISIS 814907 115 mg
Started | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 3 | 5 | 7 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 4 | 7 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0
Not completed — Voluntary Withdrawal | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator Judgement | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event or Serious Adverse Event (SAE) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Cohort A: ISIS 814907 10 mg: Participants received 10 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, Q4W on Days 1, 29, 57, and 85 in Part 1 of the study.
- Part 1: Cohort D: ISIS 814907 115 mg: Participants received 115 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, Q12W on Days 1 and 85 in Part 1 of the study.
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort A: ISIS 814907 10 mg | Part 1: Cohort B: ISIS 814907 30 mg | Part 1: Cohort C: ISIS 814907 60 mg | Part 1: Cohort D: ISIS 814907 115 mg | Part 1: Pooled Placebo | Total
Number analyzed (Participants) | 6 | 6 | 9 | 13 | 12 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (5.2) | 65.0 (6.1) | 65.6 (6.8) | 66.9 (6.3) | 66.3 (4.6) | 65.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 6 | 6 | 23
  Male | 4 | 2 | 4 | 7 | 6 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 9 | 13 | 11 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 9 | 13 | 12 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Adverse Events That Are Related to Treatment With ISIS 814907
Description: An adverse event (AE) was defined as any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of medicinal (investigational) product, whether or not the AE was considered related to the medicinal (investigational) product. A TEAE was defined as any AE that starts or worsens on or after the date of first dose of study treatment. TEAEs were categorised as mild, moderate, and severe to aid in severity assessment.
Time Frame: From first dose of study drug up to Week 37 in Part 1
Population: Safety population included all participants who were randomised and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Cohort B: ISIS 814907 30 mg: Participants received 30 mg ISIS 814907 diluted in 20 mL in artificial CSF, intrathecally Q4W on Days 1, 29, 57, and 85 in Part 1 of the study.
Arm/Group | Part 1: Cohort A: ISIS 814907 10 mg | Part 1: Cohort B: ISIS 814907 30 mg | Part 1: Cohort C: ISIS 814907 60 mg | Part 1: Cohort D: ISIS 814907 115 mg | Part 1: Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 9 | 13 | 12
Participants
  Mild | 3 | 0 | 5 | 4 | 0
  Moderate | 0 | 1 | 1 | 1 | 0
  Severe | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 2: Number of Participants With Adverse Events That Are Related to Treatment With ISIS 814907
Description: An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of medicinal (investigational) product, whether or not the AE was considered related to the medicinal (investigational) product. A TEAE was defined as any AE that starts or worsens on or after the date of first dose of study treatment. TEAEs were categorised as mild, moderate, and severe to aid in severity assessment.
Time Frame: From first dose of study drug up to Week 64 in Part 2
Population: Safety population included all participants who were randomised and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Late Start Cohort A + Cohort B + Cohort C + ISIS 814907 60 mg | Part 2: Late Start Cohort D + ISIS 814907 115 mg | Part 2: Early Start Cohort A + ISIS 814907 60 mg | Part 2: Early Start Cohort B + ISIS 814907 60 mg | Part 2: Early Start Cohort C + ISIS 814907 60 mg | Part 2: Early Start Cohort D + ISIS 814907 115 mg
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 7 | 10
Participants
  Mild | 1 | 0 | 1 | 1 | 0 | 2
  Moderate | 0 | 2 | 1 | 1 | 1 | 3
  Severe | 0 | 0 | 0 | 0 | 0 | 1

3. Secondary Outcome: CSF Trough Concentration of ISIS 814907
Time Frame: Pre dose on Day 85 in Part 1 and Day 337 in Part 2
Population: PK population consisted of all participants who were randomized, received at least 1 dose of ISIS 814907, and had sufficient sampling (at least 1 evaluable post-Baseline PK sample) to permit PK evaluation. Overall number of participants analyzed is number of participants who received active treatment (ISIS 814907) in Part 1 or received active treatment in Part 2. As pre-specified in SAP, in case of very few participants in any active treatment groups, the analysis groups may have been pooled.
Measure: Mean (Standard Deviation); unit: nanogram per millilitre (ng/mL)
Groups:
- Part 2: Cohort A + ISIS 814907 60 mg: Participants from MAD Cohort A that were ISIS 814907 10 mg-treated or placebo-treated, received 60 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, Q12W on Days 1, 85, 169, 253, and 337 in Part 2 of the study.
- Part 2: Cohort B + ISIS 814907 60 mg: Participants from MAD Cohort B that were ISIS 814907 30 mg-treated or placebo-treated, received 60 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, Q12W on Days 1, 85, 169, 253, and 337 in Part 2 of the study.
- Part 2: Cohort C + ISIS 814907 60 mg: Participants from MAD Cohort C that were ISIS 814907 60 mg-treated or placebo-treated, received 60 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, Q12W on Days 1, 85, 169, 253, and 337 in Part 2 of the study.
- Part 2: Cohort D + ISIS 814907 115 mg: Participants from MAD Cohort D that were ISIS 814907 115 mg-treated or placebo-treated, received 115 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, Q12W on Days 1, 85, 169, 253, and 337 in Part 2 of the study.
Arm/Group | Part 1: Cohort A: ISIS 814907 10 mg | Part 1: Cohort B: ISIS 814907 30 mg | Part 1: Cohort C: ISIS 814907 60 mg | Part 1: Cohort D: ISIS 814907 115 mg | Part 2: Cohort A + ISIS 814907 60 mg | Part 2: Cohort B + ISIS 814907 60 mg | Part 2: Cohort C + ISIS 814907 60 mg | Part 2: Cohort D + ISIS 814907 115 mg
Number analyzed (Participants) | 6 | 6 | 9 | 12 | 2 | 5 | 9 | 11
nanogram per millilitre (ng/mL) | 5.56 (2.12) | 9.77 (3.46) | 9.79 (3.42) | 3.26 (1.24) | 5.96 (NA) — The values were non-quantifiable [NQ] (50% of values were imputed i.e., NQ assigned zero concentration for one participant) which affected the calculation. Since only one participant had evaluable data SD was not estimable. | 8.22 (2.03) | 6.61 (2.89) | 7.82 (2.52)

4. Secondary Outcome: Maximum Observed Drug Concentration (Cmax) of ISIS 814907 in Plasma
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, and 5 hours post-intrathecal (IT) bolus injection on Day 85 in Part 1 and on Day 337 in Part 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Cohort A: ISIS 814907 10 mg | Part 1: Cohort B: ISIS 814907 30 mg | Part 1: Cohort C: ISIS 814907 60 mg | Part 1: Cohort D: ISIS 814907 115 mg | Part 2: Cohort A + ISIS 814907 60 mg | Part 2: Cohort B + ISIS 814907 60 mg | Part 2: Cohort C + ISIS 814907 60 mg | Part 2: Cohort D + ISIS 814907 115 mg
Number analyzed (Participants) | 6 | 6 | 9 | 13 | 2 | 5 | 9 | 12
ng/mL | 65.4 (203) | 285 (50.5) | 542 (148) | 830 (879) | 840 (NA) — Geometric coefficient of variation was not estimable due to insufficient number of participants with events. | 323 (56.6) | 524 (90.2) | 1011 (130)

5. Secondary Outcome: Time Taken to Reach Maximal Concentration (Tmax) of ISIS 814907 in Plasma
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, and 5 hours post-IT bolus injection on Day 85 in Part 1 and on Day 337 in Part 2
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: Cohort A: ISIS 814907 10 mg | Part 1: Cohort B: ISIS 814907 30 mg | Part 1: Cohort C: ISIS 814907 60 mg | Part 1: Cohort D: ISIS 814907 115 mg | Part 2: Cohort A + ISIS 814907 60 mg | Part 2: Cohort B + ISIS 814907 60 mg | Part 2: Cohort C + ISIS 814907 60 mg | Part 2: Cohort D + ISIS 814907 115 mg
Number analyzed (Participants) | 6 | 6 | 9 | 13 | 2 | 5 | 9 | 12
hours | 3.13 [1.02 to 24.7] | 4.00 [3.02 to 5.00] | 4.02 [2.00 to 24.2] | 3.38 [1.02 to 338] | 2.05 [1.02 to 3.08] | 4.02 [3.02 to 5.07] | 4.15 [2.02 to 24.3] | 4.03 [0.500 to 23.5]

6. Secondary Outcome: Terminal Elimination Half-life (t1/2λz) of ISIS 814907 in Plasma
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, and 5 hours post-IT bolus injection on Day 85 in Part 1 and on Day 337 in Part 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Part 1: Cohort A: ISIS 814907 10 mg | Part 1: Cohort B: ISIS 814907 30 mg | Part 1: Cohort C: ISIS 814907 60 mg | Part 1: Cohort D: ISIS 814907 115 mg | Part 2: Cohort A + ISIS 814907 60 mg | Part 2: Cohort B + ISIS 814907 60 mg | Part 2: Cohort C + ISIS 814907 60 mg | Part 2: Cohort D + ISIS 814907 115 mg
Number analyzed (Participants) | 6 | 6 | 9 | 13 | 2 | 5 | 9 | 12
days | 19.4 (62.7) | 38.0 (23.1) | 34.8 (22.6) | 42.5 (16.1) | 10.7 (NA) — Geometric coefficient of variation was not estimable due to insufficient number of participants with events. | 10.3 (8.99) | 10.6 (16.3) | 13.8 (54.0)

7. Secondary Outcome: Areas Under the Plasma Concentration-time Curve From Zero Time (Predose) to 24 Hours After the IT Administration (AUC0-24h) of ISIS 814907
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, and 5 hours post-IT bolus injection on Day 85 in Part 1 and on Day 337 in Part 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hours per millilitre (ng*h/mL)
Arm/Group | Part 1: Cohort A: ISIS 814907 10 mg | Part 1: Cohort B: ISIS 814907 30 mg | Part 1: Cohort C: ISIS 814907 60 mg | Part 1: Cohort D: ISIS 814907 115 mg | Part 2: Cohort A + ISIS 814907 60 mg | Part 2: Cohort B + ISIS 814907 60 mg | Part 2: Cohort C + ISIS 814907 60 mg | Part 2: Cohort D + ISIS 814907 115 mg
Number analyzed (Participants) | 6 | 6 | 9 | 13 | 2 | 5 | 9 | 12
nanogram*hours per millilitre (ng*h/mL) | 679 (119) | 3638 (36.0) | 6143 (92.4) | 7120 (3066) | 10523 (NA) — Geometric coefficient of variation was not estimable due to insufficient number of participants with events. | 5176 (44.5) | 6396 (68.7) | 12542 (50.2)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 37 in Part 1 and up to Week 64 in Part 2
Description: Safety population included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Part 1: Cohort D: ISIS 814907 115 mg: Participants received 115 mg ISIS 814907 diluted in 20 mL artificial CSF, intrathecally, ev(Q12W) on Days 1 and 85 in Part 1 of the study.
- Part 2: Late Start Cohort D + ISIS 814907 115 mg: Participants from MAD Cohort D that were placebo-treated, received 115 mg ISIS 814907 diluted up in 20 mL artificial CSF, Q12W on Days 1, 85, 169, 253, and 337 in Part 2 of the study.
Arm/Group | Part 1: Cohort A: ISIS 814907 10 mg | Part 1: Cohort B: ISIS 814907 30 mg | Part 1: Cohort C: ISIS 814907 60 mg | Part 1: Cohort D: ISIS 814907 115 mg | Part 1: Pooled Placebo | Part 2: Late Start Cohort A + Cohort B + Cohort C + ISIS 814907 60 mg | Part 2: Late Start Cohort D + ISIS 814907 115 mg | Part 2: Early Start Cohort A + ISIS 814907 60 mg | Part 2: Early Start Cohort B + ISIS 814907 60 mg | Part 2: Early Start Cohort C + ISIS 814907 60 mg | Part 2: Early Start Cohort D + ISIS 814907 115 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/9 | 0/13 | 0/12 | 0/4 | 0/4 | 0/3 | 0/5 | 0/7 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/9 | 0/13 | 2/12 | 1/4 | 0/4 | 1/3 | 1/5 | 0/7 | 1/10
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 9/9 | 12/13 | 9/12 | 4/4 | 3/4 | 3/3 | 4/5 | 7/7 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort A: ISIS 814907 10 mg (N=6) | Part 1: Cohort B: ISIS 814907 30 mg (N=6) | Part 1: Cohort C: ISIS 814907 60 mg (N=9) | Part 1: Cohort D: ISIS 814907 115 mg (N=13) | Part 1: Pooled Placebo (N=12) | Part 2: Late Start Cohort A + Cohort B + Cohort C + ISIS 814907 60 mg (N=4) | Part 2: Late Start Cohort D + ISIS 814907 115 mg (N=4) | Part 2: Early Start Cohort A + ISIS 814907 60 mg (N=3) | Part 2: Early Start Cohort B + ISIS 814907 60 mg (N=5) | Part 2: Early Start Cohort C + ISIS 814907 60 mg (N=7) | Part 2: Early Start Cohort D + ISIS 814907 115 mg (N=10)
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort A: ISIS 814907 10 mg (N=6) | Part 1: Cohort B: ISIS 814907 30 mg (N=6) | Part 1: Cohort C: ISIS 814907 60 mg (N=9) | Part 1: Cohort D: ISIS 814907 115 mg (N=13) | Part 1: Pooled Placebo (N=12) | Part 2: Late Start Cohort A + Cohort B + Cohort C + ISIS 814907 60 mg (N=4) | Part 2: Late Start Cohort D + ISIS 814907 115 mg (N=4) | Part 2: Early Start Cohort A + ISIS 814907 60 mg (N=3) | Part 2: Early Start Cohort B + ISIS 814907 60 mg (N=5) | Part 2: Early Start Cohort C + ISIS 814907 60 mg (N=7) | Part 2: Early Start Cohort D + ISIS 814907 115 mg (N=10)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Catheter site related reaction (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination site bruising (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrophic vulvovaginitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CSF cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Albumin CSF increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
CSF protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrophoresis protein abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haptoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transferrin saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin B12 decreased (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 3 | 1 | 2 | 3 | 3 | 0 | 1 | 0 | 0 | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 3 | 2 | 1 | 0 | 0 | 1 | 0 | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumocephalus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 3 | 2 | 3 | 1 | 0 | 1 | 1 | 1 | 4
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased vibratory sense (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Posterior cortical atrophy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 3 | 1 | 2 | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmic herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Borrelia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT03186989/Prot_SAP_000.pdf